CLINICAL TRIAL: NCT01721083
Title: Comparison of Two Methods of Immunization for Intramuscular Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: DDD# 602056
Record Dates: First submitted 2012-11-01; First posted 2012-11-05 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Consequences of Immunization Method
Keywords: intramuscular injection; bunch; z-track

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Z-Track immunization (Experimental): Subject receives Intramuscular injection by z-track method during flu vaccination given by employee health Registered Nurse into deltoid muscle.
  Interventions: Procedure: Procedure: Z-track
- Bunch immunization (Active Comparator): Subject receives Intramuscular injection by bunch method during flu vaccination given by employee health Registered Nurse into deltoid muscle.
  Interventions: Procedure: Procedure: Bunch

INTERVENTIONS:
Procedure: Procedure: Z-track — Subject received immunization by z-track
  Arms: Z-Track immunization
Procedure: Procedure: Bunch — Subject receives immunization by bunch method.
  Arms: Bunch immunization

SUMMARY:
This study is designed to compare two different styles of intramuscular injection (Bunch versus Z-Track)during flu vaccination with the following outcome measures as basis for comparison: perceive pain, redness, medication leakage, other complications within 72 hours in healthy adult volunteer subjects.

DETAILED DESCRIPTION:
This study is designed to compare two different styles of intramuscular injection (Bunch versus Z-Track)during flu vaccination with the following outcome measures as basis for comparison: perceive pain, redness, medication leakage, other complications within 72 hours in healthy adult volunteer subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults without latex allergy over 18 years of age

Exclusion Criteria:

* latex allergy
* illness
* 18 years or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Perceived pain | 72 hours
  Subjects will be asked to rate perceived pain on scale of 0-10

SECONDARY OUTCOMES:
Medication leakage | 72 hours
  Any medication leakage from either arm within 72 hours
Redness at injection site | 72 hours
  Redness, as determined by naive observer at injection site immediately and up to 72 hours after study.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E Bayne, PhD, ARNP, NNP-BC, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States